CLINICAL TRIAL: NCT01265407
Title: Malaria Surveillance in Rakai, Uganda
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911050; 11-I-N050
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Malaria
Keywords: Children; Hemoglobinopathies; Epidemiology; Natural History; Malaria
MeSH Terms: conditions — Malaria; Hemoglobinopathies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

- Malaria is a leading cause of morbidity and mortality in Uganda, accounting for more than a quarter of all outpatient visits at health facilities, 20 percent of hospital admissions, and about 10 percent of inpatient deaths. Children under 10 years of age, pregnant women, and HIV-infected individuals bear the greatest burden of disease. To provide baseline information for future malaria vaccine research, development, and testing, researchers are interested in collecting malaria infection data from the Rakai district in southern Uganda.

Objectives:

- To assess the epidemiology of malaria infection among children aged 6 months to less than 10 years and adults living in same households with children in Rakai district, Uganda.

Eligibility:

- Children between 6 months and 10 years of age, as well as their primary caregiver and an additional randomly selected adolescent or adult resident of the household, from the Rakai district of Uganda.

Design:

* Participants will have monthly household visits for a 1-year surveillance period.
* Each visit will include a structured interview/questionnaire of the primary caregiver or legal guardian of the child and clinical and laboratory assessments of each child, the primary caregiver, and the additional adolescent or adult resident of the household. The questionnaire will ask about malaria treatment and prevention measures.
* Children will provide a blood sample for testing. Individuals (children or adults) who are diagnosed with malaria or anemia during the course of the study will be recommended for treatment.
* Researchers will also track usage of the district health clinic and hospital services to link medical records for study participants.

DETAILED DESCRIPTION:
Malaria is a leading cause of morbidity and mortality in Uganda, accounting for 25-40 percent of all outpatient visits at health facilities, 20 percent of hospital admissions, and 9-14 percent of inpatient deaths. Malaria is meso- to holoendemic in Rakai, southwestern Uganda and children under 10 years, pregnant women and HIVinfected individuals bear the greatest burden of disease. Substantial progress has been made in malaria vaccine development and vaccine trials will be conducted over the coming years. The design of these trials will be contingent on understanding the epidemiology of malaria and disease burden in different epidemic settings.

This study will determine the epidemiology of malaria infection in children and adolescents/adults by conducting surveillance in approximately 320 households selected from two of the 10 clusters under the Rakai Community Cohort Study (RCCS). Monthly visits will be made to randomly selected households during a one year surveillance period. Visit procedures include: structured interview/questionnaire of the primary care giver or legal guardian of the child; clinical and laboratory assessment of each child aged 6 months up to 10 years and the primary care giver; and clinical and laboratory assessment of one additional randomly selected adolescent/adult resident of the household. The study team will track usage of health clinic or hospital services within the district in order to link medical records for study participants. This community-based surveillance study will be linked to a separate facility-based surveillance study in health clinics/hospitals servicing the selected communities. This study will enhance the investigators understanding of the epidemiology of pediatric and adult malaria infection in Rakai district in preparation for future malaria vaccine trials. Investigators will be able to estimate the incidence of uncomplicated and severe malaria in children and adults. This protocol will also investigate the prevalence and association of sickle cell trait, xlinked glucose-6-phosphatase dehydrogenase deficiency and hemoglobinopathies (Hemoglobin C) and their associations with severe malaria among children and adults.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Child aged 6 months to less than 10 years, primary care giver of an enrolled child, or an adolescent/adult resident in a household of an enrolled child.
  2. Willingness to participate in the study as evidenced by a completed and signed parental informed consent document and consent for child research participation (with assent of child/adolescent if appropriate).

EXCLUSION CRITERIA:

1. Clinical evidence of an acute, life-threatening illness requiring immediate medical care at time of baseline household visit, not including severe malaria.
2. Intent to stay in a study household for less than 12 months from the start of the study.
3. School-going child in a boarding school who spends most of their time in a year at school rather than at home.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1600 participants in approximately 320 households.@@@N=1700
Sampling Method: Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2010-12-22 (Actual); Primary Completion 2012-09-12 (Actual); Study Completion 2013-07-23 (Actual)

PRIMARY OUTCOMES:
Episodes of uncomplicated and severe clinical malaria per year in children and adults. | 1 year
  to assess the epidemiology of malaria infection among children aged 6months-1year and adults living in the same household with children in Rakai district

SECONDARY OUTCOMES:
Malaria rates (episodes/per year) in individuals and communities and by seasonality. Clinical episodes will be determined using RDT among febrile participants. | 1 year
  to estimate the proportion of participants from the household surveillance that seek care for malaria in health facilities
Determine the rates of asymptomatic parasitemia among afebrileparticipants (determined by malaria smears and PCR). | 1 year
  to coordinate the community based surveillance with a facility based surveillance in health clinics servicing the selected communities
The prevalence of enlarged palpable spleen (splenomegaly) in children | 1 year
  to investigate the prevalence of sickle cell trait,glucose-6 phosphate dehydrogenase deficiency and hemoglobinopathies and their relationship to severe clinical malaria per year in children and adults.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Rakai Health Sciences Program, Rakai, Uganda

REFERENCES:
- [Background] Hopkins H, Bebell L, Kambale W, Dokomajilar C, Rosenthal PJ, Dorsey G. Rapid diagnostic tests for malaria at sites of varying transmission intensity in Uganda. J Infect Dis. 2008 Feb 15;197(4):510-8. doi: 10.1086/526502. PMID 18240951
- [Background] Jensen TP, Bukirwa H, Njama-Meya D, Francis D, Kamya MR, Rosenthal PJ, Dorsey G. Use of the slide positivity rate to estimate changes in malaria incidence in a cohort of Ugandan children. Malar J. 2009 Sep 15;8:213. doi: 10.1186/1475-2875-8-213. PMID 19754955
- [Background] Pullan RL, Bukirwa H, Staedke SG, Snow RW, Brooker S. Plasmodium infection and its risk factors in eastern Uganda. Malar J. 2010 Jan 4;9:2. doi: 10.1186/1475-2875-9-2. PMID 20044942
- [Derived] Newell K, Kiggundu V, Ouma J, Baghendage E, Kiwanuka N, Gray R, Serwadda D, Hobbs CV, Healy SA, Quinn TC, Reynolds SJ. Longitudinal household surveillance for malaria in Rakai, Uganda. Malar J. 2016 Feb 9;15:77. doi: 10.1186/s12936-016-1128-6. PMID 26861943